CLINICAL TRIAL: NCT03326089
Title: Short and Long-term Effects of Oxygen Supplemented Pulmonary Rehabilitation in Idiopathic Pulmonary Fibrosis
Brief Title: Pulmonary Rehabilitation in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corfu General Hospital (Other)
Responsible Party: Principal Investigator, Ilias Papanikolaou, Consultant Pulmonary Physician, Corfu General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CorfuGH569
Record Dates: First submitted 2017-10-17; First posted 2017-10-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: pulmonary rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: participants are blindly randomized to receive oxygen or not during rehabilitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow oxygen supplementation (Active Comparator): Pulmonary rehabilitation with constant high flow supplementary oxygen supply FiO2 50% for 2 months (Group A).
  Interventions: Procedure: Pulmonary rehabilitation
- Oxygen supplementation upon hypoxemia (Placebo Comparator): Pulmonary rehabilitation without oxygen supply unless upon resting or exercise induced hypoxemia for 2 months (Group B).
  Interventions: Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — Endurance training for 30 minutes, 3 times/week for 2 months followed by resistance training
  Other Names: oxygen supplementation

SUMMARY:
This is an interventional double-blind randomized controlled trial, to investigate the short and long-term effects of a supervised exercise training program in patients with IPF, depending on alternate patterns of oxygen supplementation during PR.

DETAILED DESCRIPTION:
The investigators hypothesize that PR service with supplemented oxygen supply regardless of hypoxemia may have significantly better short-term effects in patients with IPF. The study will take place in Corfu General Hospital, by the Departments of Pulmonary Medicine and Physiotherapy and Rehabilitation, respectively. Study participants will be divided in two equal arms 1:1 in a double-blind manner. One of the investigators blinded to their clinical data will assign each participant to PR service either i) with constant supplementary oxygen supply FiO2 50% regardless of saturation status Group A) or ii) without oxygen supply unless upon resting or exercise induced hypoxemia (saturation <88%) (Group B).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IPF based on current established criteria
* no exacerbation previous 3 months
* no participation in such program previous 3 months.
* If on treatment with pirfenidone or nintedanib, this will be recorded and patient should be on treatment for at least 3-6 months to achieve stable state.

Exclusion Criteria:

- concomitant diagnosis of congestive heart failure and lung cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test Distance (6MWTD) (meters) | 2 months
  Statistically significant short term effect on exercise capacity
Saint-George Respiratory Questionnaire Idiopathic Pulmonary Fibrosis Version (SGRQ-I) (units on scale) | 2 months
  Statistically significant short term effect on health related quality of life
Hospital Anxiety and Depression Scale (HADS) (units on scale) | 2 months
  Statistically significant short term effect on health related quality of life

SECONDARY OUTCOMES:
6 Minute Walk Test Distance (6MWTD) (meters) | 12 months
  Statistically significant long term effect on exercise capacity
Saint-George Respiratory Questionnaire Idiopathic Pulmonary Fibrosis Version (SGRQ-I) (units on scale) | 12 months
  Statistically significant long term effect on health related quality of life
Hospital Anxiety and Depression Scale (HADS) (units on scale) | 12 months
  Statistically significant long term effect on health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Stefanos Patsiris, Study Director — Physiotherapy Director
Locations (1):
- Corfu General Hospital, Corfu, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Everything will be published in time.